CLINICAL TRIAL: NCT06449300
Title: Effects of Different Volumes of Resistance Training on Body Composition, Peak Power, and Muscle Thickness in Untrained Healthy Women
Brief Title: Effects of Different Volumes of Resistance Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Princess Nourah Bint Abdulrahman University (Other)
Collaborators: Kırıkkale University (Other)
Responsible Party: Principal Investigator, Monira Aldhahi, Associate professor, Princess Nourah Bint Abdulrahman University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021.11.07
Record Dates: First submitted 2024-06-01; First posted 2024-06-10 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Healthy
Keywords: Strength training; muscle growth

STUDY DESIGN:
Who Masked: Investigator
Masking Description: a researcher blinded to the interventions
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- low volume (LVT) resistance training (Experimental): 3 sessions of 12 exercises per week for 8 weeks . Split-strength training method will be applied. After participants' 1RM maximums were determined, training loads were calculated separately for each participant. All workouts will be conducted by certified trainers to ensure they are performed in the correct training format. Each training session lasted approximately 60 minutes. The weekly training loads of all participants will be increased by 5%. In the MVT group, 3 sets of 8-12 repetitions: between sets intervals: of 120 seconds will be performed.
  Interventions: Other: Resistance exercise-LVT
- moderate volume (MVT) resistance training (Active Comparator): 4 sessions of 12 exercises per week for 8 weeks . Split-strength training method will be applied. After participants' 1RM maximums were determined, training loads were calculated separately for each participant. All workouts will be conducted by certified trainers to ensure they are performed in the correct training format. Each training session lasted approximately 60 minutes. The weekly training loads of all participants will be increased by 5%. In the MVT group, 3 sets of 8-12 repetitions: between sets intervals: of 120 seconds will be performed.
  Interventions: Other: Resistance exercise-MVT
- high volume (HVT) resistance training (Active Comparator): 5 sessions of 12 exercises per week for 8 weeks . Split-strength training method will be applied. After participants' 1RM maximums were determined, training loads were calculated separately for each participant. All workouts will be conducted by certified trainers to ensure they are performed in the correct training format. Each training session lasted approximately 60 minutes. The weekly training loads of all participants will be increased by 5%. In the MVT group, 3 sets of 8-12 repetitions: between sets intervals: of 120 seconds will be performed.
  Interventions: Other: Resistance exercise-HVT

INTERVENTIONS:
Other: Resistance exercise-LVT — (low volume training - 3 sessions of 12 exercises per week)
  Arms: low volume (LVT) resistance training
Other: Resistance exercise-MVT — (moderate volume training - 4 sessions of 12 exercises per week)
  Arms: moderate volume (MVT) resistance training
Other: Resistance exercise-HVT — (high volume training - 5 sessions of 12 exercises per week)
  Arms: high volume (HVT) resistance training

SUMMARY:
This study explores the effects of varying volumes of resistance training on body composition, strength, peak power, and muscle thickness in untrained women over eight weeks. A randomized controlled trial involving 45 female college students assessed the outcomes across three groups: low-volume training (LVT) with three weekly sessions, moderate-volume training (MVT) with four weekly sessions, and high-volume training (HVT) with five weekly sessions. Participants were untrained, aged 18-65, and free from cardiovascular diseases or performance-enhancing drugs.

The hypothesis suggested that moderate volume training would yield optimal muscle development, considering the potential non-linear dose-response relationship where excessive training might be detrimental. Measurements included body composition, muscle thickness, and peak power through a force platform during vertical jumps.

Data analysis focused on changes in muscle thickness, strength, and body composition, with statistical significance set at p < 0.05. The study aimed to provide insights into how different training volumes affect physiological adaptations in untrained women, potentially guiding fitness regimen optimizations for similar populations.

DETAILED DESCRIPTION:
The study aimed to investigate the effect of different resistance training volume (low-, moderate, and high) on body composition, maximal strength, peak power, and muscle thickness in untrained women over eight weeks. The study is a three-arm, randomized controlled trial, 45 female college students participated, fit the specific inclusion criteria like age between 18-65 and being untrained. Exclusion criteria included the use of performance-enhancing drugs or recent resistance training.

Participants were randomly assigned to one of three groups: low-volume training (LVT) with three sessions weekly, moderate-volume training (MVT) with four sessions weekly, and high-volume training (HVT) with five sessions weekly. Each session comprised 12 exercises. Split split-strength training method was applied. After participants' 1RM maximums were determined, training loads were calculated separately for each participant. All workouts were conducted by certified trainers to ensure they were performed in the correct training format. Each training session lasted approximately 60 minutes. The weekly training loads of all participants were increased by 5%. In the LVT group, 3 sets of 8-12 repetitions of: between sets interval: 120 seconds (3 days/wk), in the MVT group, 3 sets of 8-12 repetitions of: between sets interval: 120 seconds (4 days/wk), in the HVT group, 3 sets of 8-12 repetitions of: between sets interval: 120 seconds exercises (5 days/wk) were performed.

Results and data analysis involved anthropometric measurements, muscle thickness via ultrasound, and peak power from the vertical jump test. Statistical significance was set at p < 0.05, and effect sizes were calculated with Partial Eta Squared values.

ELIGIBILITY:
Inclusion Criteria:

* Adult women between ages of 18 -65 years old
* Able to walk independently
* Free of any history of cardiovascular disease
* Untrained (less than 150 min of PA/week)

Exclusion Criteria:

* Intake of performance-enhancing drugs, anabolic steroids
* Any history of injury, or physiological or physical limitations that could affect the ability to perform training and physical testing in the last year.
* Those who had been RT for more than 2 months in the previous 6 months were excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-11-11 (Actual); Primary Completion 2023-12-11 (Actual); Study Completion 2024-01-11 (Actual)

PRIMARY OUTCOMES:
Body height measurements | at baseline and end of 8 week
  A stadiometer is attached to the wall. It has a sliding horizontal headpiece that's adjusted to rest on top of your head. The measurement of height will be conducted using a Mesilife portable stadiometer.
Anthropometric measurements | at baseline and end of 8 week
  Bio-impedance body composition analysis system
Muscle thickness measurements | at baseline and end of 8 week
  A portable ultrasound scanner will be used to determine muscle thickness. At one location, muscle thickness will be measured: Between the greater trochanter and the lateral epicondyle of the thigh, the thickness of the quadriceps femoris (Vastus lateralis) will be measured at 50%. Ultrasound tests will be done at the start of the study and 8 weeks later, by a researcher blinded to the interventions. All tests were performed in the morning when participants are fasting.
Countermovement Jump (CMJ) | at baseline and end of 8 week
  Countermovement Jump (CMJ) values of all participants will be measured. Peak muscle power measures in watts (W) using the Accupeak power2.0 portable force platform system . The measurement frequency of the device was set to 500 Hz. Participants will undrergo a 10-minute warm-up program before completing a CMJ. Participants will be asked to begin a downward movement and jump as high as possible after hearing a tone from the computer.

CONTACTS AND LOCATIONS:
Overall Officials: Dondu Ugurlu, Phd, Principal Investigator — dondusimsek@kku.edu.tr
Locations (1):
- Princess Nourah bint Abdulrahman University, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ugurlu D, Gulu M, Yapici H, Yagin FH, Comertpay E, Eroglu O, Afonso J, Aldhahi MI. Dose-response effects of 8-week resistance training on body composition and muscular performance in untrained young women: A quasi-experimental design. Medicine (Baltimore). 2024 Nov 1;103(44):e40322. doi: 10.1097/MD.0000000000040322. PMID 39496043